CLINICAL TRIAL: NCT05859425
Title: Investigation of Real-time Diagnostic Ultrasound as a Means of Biofeedback Training in Transversus Abdominus Re-education of Patients With Non-specific Low Back Pain: Prospective Randomized Controlled Pilot Study
Brief Title: Ultrasound-guided Biofeedback for Transversus Abdominus Re-education in Non-specific Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Collaborators: University of Crete (Other)
Responsible Party: Principal Investigator, Evdokia Billis, Professor in Physiotherapy, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Non-specific Low Back Pain (NSLBP)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided biofeedback intervention (Experimental): This group received visual feedback using real-time ultrasound (US) for transversus abdominus (TrA) activation, while performing the exercise programme. US-guided TrA imaging was initially performed with participants in crook lying, with the US head positioned along the lateral abdominal wall with reference points at the lower point of the rib cage (last rib) and the anterior superior iliac spine, on the right side of the person, midway between these two points. The US head was moved until the user (health professional-investigator) had the best possible visualization of the lateral abdominal muscles (external oblique, internal oblique and TrA). During the execution of the exercises, the participants could watch the ultrasound screen along with the therapist's guidance, thus receiving information (US-visual feedback) of their TrA activation.
  Interventions: Device: Real-time rehabilitative ultrasound imaging (RUSI)
- Control (non-US guided) group (Active Comparator): The control group received the traditional tactile feedback from the therapist while performing the motor control exercises for TrA activation. Traditionally, assessment of TrA contraction involves palpation of the muscles. The ability to assess TrA through muscle palpation is largely dependent on examiner's skill, as TrA cannot be directly palpated (feedback sensation being limited from internal oblique muscle). To control the activation of the abdominals the therapist placed his hands on the inside of the anterior superior iliac crests (tactile feedback) and instructed the examinee to pull the abdominal wall inward without moving the spine or pelvis (verbal feedback). The same exercise protocol to the experimental group was performed in this (control) group.
  Interventions: Other: Tactile feedback (control intervention)

INTERVENTIONS:
Device: Real-time rehabilitative ultrasound imaging (RUSI) — Τhe ultrasound equipment used was B-K Μedical Mini Focus 1402 equipped with high frequency linear probe (8670, 5-12MHz) using standard musculoskeletal settings and the software: V 1.01.01.137. Ultrasound gel (AQUASONIC® 100, Parker Inc., Orange, NJ) was used as coupling agent. TrA imaging was initially performed with participants in crook lying, with the US head positioned along the lateral abdominal wall with reference points at the lower point of the rib cage (last rib) and the anterior superior iliac spine, on the right side of the person, midway between these two points. The US head was moved until tester (investigator) had the best possible visualization of the lateral abdominal muscles (external oblique, internal oblique and TrA). During the execution of the exercises, the participants could watch the ultrasound screen along with the therapist's guidance, thus receiving information (US-visual feedback) of their TrA activation
  Arms: US-guided biofeedback intervention
Other: Tactile feedback (control intervention) — Palpatory-guided (manual) feedback for TrA activation
  Arms: Control (non-US guided) group

SUMMARY:
As rehabilitative ultrasound imaging (RUSI) for monitoring and re-educating deep trunk muscles is becoming more and more popular in current musculoskeletal rehabilitation and research, the purpose of this pilot study was to explore the effects of applying ultrasound-guided imaging as a means of feedback for the activation/contraction of the deep transervsus abdominis muscle of the trunk during an exercise programme in people with non-specific low back pain (NSLBP). The outcome mesures being explored were pain intensity (primary outcome) through Numeric Pain Rating Scale (NPRS), functional, muscular and psychosocial parameters.

DETAILED DESCRIPTION:
Background: It is believed that ultrasound-guided imaging of activation/contraction of the deep abdominal muscles (such as transervsus abdominis) is useful for assisting deep muscle re-education, which is often dysfunctional in non-specific low back pain (NSLBP). Thus, this pilot study aimed to evaluate the use of real-time ultrasound (US) as a feedback device for transverse abdominis (TrA) activation/contraction during an exercise program in chronic NSLBP patients.

Methods: Chronic NSLBP patients are recruited and randomly assigned to an US-guided or control group. The same motor control-based exercise program is applied to both groups. All patients would receive physiotherapy twice per week for 7 weeks. Outcome measures, tested at baseline and post-intervention, include Numeric Pain Rating Scale (NPRS), TrA activation level (measured through a pressure biofeedback unit-based developed protocol), seven established motor control tests, Roland-Morris Disability Questionnaire (RMDQ) and Hospital Anxiety and Depression Scale (HADS). Analysis of variance utilizing a two-way mixed ANOVA model for dependent measures of two factors (treatment group and time point of measurement) of which only one is repeated (time point of measurement) is performed to determine between- and within-group differences before and after treatment. Additionally, independent samples' t-test and paired samples' t-test are used for differences between and within groups, respectively, as well as χ2 tests for differences on the motor control tests and the TrA activation level procedure across the groups.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-60 years-old
* suffered from NSLBP lasting longer than 12 weeks, producing moderate or severe disability

Exclusion Criteria:

* people with previous spinal surgery
* people suffering from systemic diseases
* pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Change from baseline Numeric Pain Rating Scale at 2 months
  Pain intensity measure, in a 0-10 point scale, where 0 refers to NO PAIN and 10 to the WORST PAIN

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMDQ) | Change from baseline Roland Morris Disability Questionannaire at 2 months
  Disability measure, in a 0-24 point scale, where 0 refers to no disability and 10 to severe disability
Hospital Anxiety and Depression Scale (HADS) | Change from baseline Hospital Anxiety and Depression Scale at 2 months
  Anxiety and Depression scale, measuring Anxiety and Depresion. Each subscale is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression.
Transversus Abdominus (TrA) Activation Level | Change from the baseline Transversus abdominus activation level at 2 months
  Muscular assessment for evaluating TrA activation level using the stabilizer pressure biofeedback unit (Chattanooga Group model, US) was developed and tested for its reliability for the purposes of this study. The activation levels for allowing exercise progressions to take place were determined (categorically) as follows: Level 1: Single contraction of the TrA, lasting 10sec Level 2: Three TrA abdominal contractions, lasting 10sec Level 3: Ten abdominal TrA contractions, lasting 10sec Level 4: Holding the TrA contraction while performing 5 repetitions of side bend-ing (and return) of each leg (bend knee fallout and return) Level 5: Holding the TrA contraction while performing 5 bend leg raises on each leg Level 6: Holding the TrA contraction while performing 5 repetitions of bending and extending each leg (leg slides).
Motor Control Tests (MCT) | Change from the baseline motor control tests (how many performed CORRECTLY) at 2 months
  7 lumbopelvic clinical tests for assessming control of movement (marked as CORRECT or INCORRECT -nominal type data) Seven reliable motor control tests previously utilized with chronic NSLBP populations. These were: i) waiters bow, ii) pelvic tilt, iii) hook lying position, iv) quadruped position (flexion-control), v) quadruped position (exten-sion-control), vi) prone lying active knee flexion and vii) sitting knee extension. An in-ter-tester reliability procedure for these tests was conducted prior to data collection. Physiotherapists (testers) visually evaluated the movement quality of these tests, marked as correct or incorrect, as indicated in relevant literature.

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, Principal Investigator — University of Patras
Locations (1):
- Laboratory of Clinical Rehabilitation and Research, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we think we would be happy to proceed further and then make data publicly available.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05859425/Prot_SAP_000.pdf